CLINICAL TRIAL: NCT06973967
Title: Evaluation of the Association Between Low-Flow and Normal-Flow Anesthesia and Postoperative Delirium in Elderly Patients Undergoing Hip Fracture Surgery
Brief Title: Low- vs. Normal-Flow Anesthesia and Delirium After Hip Fracture in the Elderly
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, veysel Dinç, Assist. Prof., Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH, VD
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Delirium - Postoperative; Low Flow Anesthesia; Elderly Patients (>65 Years); Hip Surgery
Keywords: delirium; hip surgery; elderly patients; low-flow anesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients over the age of 65 who undergo hip fracture surgery under general anesthesia: Patients over the age of 65 who undergo hip fracture surgery under general anesthesia
  Interventions: Behavioral: delirium

INTERVENTIONS:
Behavioral: delirium — Postoperatively, patients were monitored for delirium for seven days.

SUMMARY:
The aim of this study is to investigate the relationship between low-flow and normal-flow anesthesia techniques and the development of postoperative delirium in elderly patients undergoing surgery for hip fracture.

DETAILED DESCRIPTION:
Materials and Methods:

Study Design and Ethical Approval:

This study is designed as a prospective observational study. Ethical approval has been obtained, and the study will be conducted in accordance with the principles of the Declaration of Helsinki. Written informed consent will be obtained from all patients enrolled in the study.

There will be no intervention or randomization by the investigators in the selection of patients; the choice between low-flow and normal-flow anesthesia will be left to the discretion of the attending anesthesiologist as per routine clinical practice. Patients aged ≥65 years who are admitted to SBÜ Gaziosmanpaşa Training and Research Hospital due to hip fracture and are scheduled for surgery will be included in the study.

This is a single-center study. Postoperative outcomes including the incidence and duration of delirium on postoperative days 1, 3, and 7, visual pain and sedation scores, length of hospital stay, and associated complications will be evaluated. Postoperative sedation will be assessed using the Richmond Agitation-Sedation Scale (RASS), and pain will be assessed using the Visual Analog Scale (VAS), both of which are part of routine hospital practice. In addition, the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) will be used to evaluate the presence of delirium in study participants.

The study is planned to continue for a duration of six (6) months.

Study Population:

Inclusion Criteria:

Patients aged 65 years and older who are scheduled to undergo surgical treatment for hip fracture, classified as ASA physical status I-IV, and who have signed the informed consent form will be included in the study.

Exclusion Criteria:

Patients with complex fractures (multiple fractures, extremity, abdominal, pelvic or sacral trauma, head trauma, etc.), those with relative contraindications to general anesthesia (e.g., known difficult airway, malignant hyperthermia), patients requiring postoperative intubated intensive care follow-up, those with a history of dementia, sleep disorders, or psychosis, individuals with serious neurological diseases (e.g., Parkinson's disease, stroke sequelae), those with a history of opioid, alcohol, or substance use, patients with cerebrovascular disease, those who underwent surgery within the past 6 months, patients with hearing or vision impairment, bleeding disorders or those taking medications affecting coagulation, patients with hypoalbuminemia (<3 g/dL), preoperative anemia with hematocrit <30%, known allergy to anesthetic drugs, severe cardiopulmonary failure, immobility, malnutrition, or those who are unable to comply with the study protocol will be excluded from the study.

Data Collection:

Demographic data of the patients (age, gender, body mass index, and comorbidities) as well as their preoperative cognitive status will be recorded. During the perioperative period, data including vital parameters, medications used, duration of anesthesia, amount of blood loss, and fluid balance will be collected.

Postoperative Assessment:

Postoperative delirium will be assessed on postoperative days 1, 3, and 7 using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), the Visual Analog Scale (VAS), and the Richmond Agitation-Sedation Scale (RASS). In addition, intensive care unit (ICU) requirement, length of hospital stay, and mortality rates of the patients will be recorded.

Statistical Methods to Be Used:

• The data will be analyzed using SPSS version 25.0 (IBM Company).

Analysis of Demographic and Clinical Data:

* Frequency and percentage distributions will be calculated for categorical variables such as patients' demographic characteristics, smoking and alcohol use, type and amount of analgesics, use of blood products, amount of bleeding, presence of chronic diseases, height, weight, body mass index (BMI), duration of surgery, length of hospital stay, and anesthesia techniques.
* To examine the relationships between categorical variables, the Chi-square test or Fisher's exact test will be used as appropriate. The independent samples t-test will be applied where necessary. Correlation or regression analysis will be used to examine the relationships between numerical variables. The statistical significance of differences will be evaluated using the Log-rank test.

Optimization Techniques (Minitab):

• If needed, optimization techniques such as Response Surface Methodology (RSM) may be applied using the Minitab statistical software.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 65 years and older who are scheduled to undergo surgical treatment for hip fracture, classified as ASA physical status I-IV, and who have signed the informed consent form will be included in the study.

Exclusion Criteria:

Patients with complex fractures (multiple fractures, extremity, abdominal, pelvic or sacral trauma, head trauma, etc.), those with relative contraindications to general anesthesia (e.g., known difficult airway, malignant hyperthermia), patients requiring postoperative intubated intensive care follow-up, those with a history of dementia, sleep disorders, or psychosis, individuals with serious neurological diseases (e.g., Parkinson's disease, stroke sequelae), those with a history of opioid, alcohol, or substance use, patients with cerebrovascular disease, those who underwent surgery within the past 6 months, patients with hearing or vision impairment, bleeding disorders or those taking medications affecting coagulation, patients with hypoalbuminemia (<3 g/dL), preoperative anemia with hematocrit <30%, known allergy to anesthetic drugs, severe cardiopulmonary failure, immobility, malnutrition, or those who are unable to comply with the study protocol will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly Patients Undergoing Hip Fracture Surgery
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium is lower in patients receiving low-flow anesthesia compared to those receiving normal-flow anesthesia. | 7 days

SECONDARY OUTCOMES:
28-day mortality | 28 days
Correlation Between NIRS Monitoring Values and Postoperative Delirium | 7 days
  Postoperative delirium will be assessed using the Confusion Assessment Method for the ICU (CAM-ICU). NIRS will be recorded intraoperatively as mean regional cerebral oxygen saturation (%). Correlation between mean NIRS values and the incidence of postoperative delirium will be analyzed.
Correlation Between BIS Values and Postoperative Delirium | First 7 postoperative days
  BIS values (mean intraoperative BIS score) will be recorded and correlated with postoperative delirium status measured by CAM-ICU.

IPD SHARING:
Plan to Share IPD: No